CLINICAL TRIAL: NCT03185156
Title: The Preventive Effect of Sub Hypnotic Dose of Propofol for Nausea and Vomiting Induced by Hemabate
Brief Title: The Preventive Effects of Sub Hypnotic Dose of Propofol for Nausea and Vomiting Induced by Hemabate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Yanmei-Bi, Principal Investigator, West China Second University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WESTCHINASUHA-023
Record Dates: First submitted 2017-06-10; First posted 2017-06-14 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Nausea and Vomiting
Keywords: nausea and vomiting; hemabate; propofol
MeSH Terms: conditions — Nausea; Vomiting | interventions — Propofol; Saline Solution

STUDY DESIGN:
Intervention Model Description: 60 maternal aged 20-40 years will be collected
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol group (Experimental): first dose 0.3mg/Kg propofol, then 1mg/Kg/hr micro-pump
  Interventions: Drug: Propofol
- control group (Placebo Comparator): first dose 0.03ml/Kg normal saline, then 0.1ml/Kg/hr micro-pump
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Propofol — first dose 0.3mg/Kg propofol, then 1mg/Kg/hr micro-pump
  Arms: propofol group
Drug: Normal saline — first dose 0.03ml/Kg placebo saline, then 0.1ml/Kg/hr micro-pump
  Arms: control group

SUMMARY:
This is a randomized, placebo-controlled trail, the objective of this study is observation the effect of sub hypnotic dose of propofol for prevention of nausea and vomiting induced by hemabate during spinal anesthesia for elective cesarean section. The primary outcome is the presence of post-delivery intra-operative nausea and vomiting in parturients. The patients demographic characteristics, blood pressure, sensory block level, and the medications will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-40 years;
* American Standards Association status I-II.

Exclusion Criteria:

* Patients with allergy or hypersensitivity to propofol, lipid emulsion, or granisetron;
* History of nausea or vomiting within 24h before cesarean delivery;
* History of gastrointestinal or psychiatric disease, motion sickness, smoking, postoperative nausea and vomiting;
* Morbid obesity;
* Consumption of drugs such as opioids, antiemetics , H2 antagonists, phenothiazines and/or corticosteroids within 24h before the study period;
* Any chronic medical or surgical disorders complicating the pregnancy;
* Conditions contraindicating regional anesthesia.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
The presence of nausea and vomiting | 24 hours
  the patients were not asked directly about nausea during the course of the surgery, but its incidence was recorded when spontaneously reported vomiting was recorded as observed by investigator

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
published in paper form
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Bi Y, Zhong R, Huang J, Huang H. Effect of continuous infusion of a subhypnotic dose of propofol on nausea and vomiting after carboprost administration at cesarean delivery: A randomized, double-blind, placebo-controlled trial. Int J Gynaecol Obstet. 2022 May;157(2):283-288. doi: 10.1002/ijgo.13742. Epub 2021 Jun 9. PMID 33993473